CLINICAL TRIAL: NCT06207357
Title: Optical Trocar to Facilitate the Pneumoperitoneum Creation in Bariatric Patients: Our Experience and Systematic Review
Brief Title: Optical Trocar to Create the Pneumoperitoneum in Bariatric Patients
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Giovanna Pavone, Medical doctor, University of Foggia
Other Study IDs: 9
Record Dates: First submitted 2023-12-15; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate; Surgery-Complications
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: optical trocar to create the pneumoperitoneum for bariatric surgery — The technique involves the use of 4 12 mm trocars. Pneumoperitoneum is induced by a 0° optical trocar and maintained at 15 mmHg. The first trocar is usually inserted along the left mid-clavicular line approximately 2 fingers from the costal arch, another trocar along the left axillary line, a third trocar 1 cm to the right of the midline, and the fourth trocar along the right mid-clavicular line. A 10 mm, 30 ° laparoscope is used.

SUMMARY:
Laparoscopic bariatric surgery are becoming the most used procedure to treat the obesity. To facilitate safe initial access to the abdominal cavity, we insert an optical viewing trocar at the left hypocondrium. The aim of this study is to systematically evaluate all published data existing in the literature to analyze the safety of optical trocars in patients undergoing bariatric surgery and to compare these data with our experiences.

DETAILED DESCRIPTION:
In this study we analyze data existing in the literature about the use of the optical trocars in patients undergoing bariatric surgery and we compare these data with our experiences.

Establishing pneumoperitoneum is classically performed using a Veress needle or the open Hasson technique, but obesity presents its own challenges when using these techniques, including thickened abdominal wall, variable anatomical landmarks, difficult and time-consuming dissection, air leak, inadequate pneumoperitoneum, subcutaneous emphysema, and difficulty with fascial closure

ELIGIBILITY:
Inclusion Criteria:

BMI>40 kg/m2 BMI>35 kg/m2with at least one associated major comorbidity

Exclusion Criteria:

secondary obesity due to endocrine and psychological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Body mass index (BMI) ≥35-39 kg/m2 with one obesity- associated co-morbidity or BMI≥40kg/m2, age ≥ 18 years.
Sampling Method: Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
optical trocar to induce the pneumoperitoneum | 5 years
  the use of optical trocar to facilitate the creation of the pneumoperitoneum in obese patients underwent bariatric surgery
complication rate using optical trocar to create the pneumopritoneum in laparoscopic surgery | 5 years
  in literature we observe a low complication rate which include bowel and vessel injuries

CONTACTS AND LOCATIONS:
Locations (1):
- Giovanna Pavone, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT06207357/Prot_000.pdf